CLINICAL TRIAL: NCT02481128
Title: Randomized Controlled Multicenter Surgical Trial to Evaluate the Impact of a Lymphoscintigraphy Prior to Sentinel Node Biopsy in Early Breast Cancer; SenSzi (GBG80)
Brief Title: Surgical Trial to Evaluate the Impact of a Lymphoscintigraphy Prior to Sentinel Node Biopsy in Early Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kliniken Essen-Mitte (Other)
Collaborators: GBG Forschungs GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SenSzi (GBG80)
Record Dates: First submitted 2015-06-05; First posted 2015-06-25 (Estimated); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Early-Stage Breast Carcinoma
Keywords: lymphoscintigraphy; sentinel lymph node biopsy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (access to lymphoscintigraphy) (No Intervention): Axillary sentinel lymph node biopsy with preoperative access to lymphoscintigraphy findings
- B (no access to lymphoscintigraphy) (Experimental): Axillary sentinel lymph node biopsy without preoperative access to lymphoscintigraphy findings
  Interventions: Procedure: without preoperative access to lymphoscintigraphy findings

INTERVENTIONS:
Procedure: without preoperative access to lymphoscintigraphy findings — axillary sentinel lymph node biopsy without access to lymphoscintigraphy findings
  Arms: B (no access to lymphoscintigraphy)

SUMMARY:
Sentinel node biopsy is a well established tool for axillary staging in early breast cancer. So far the impact of a preoperative lymph node scintigraphy is unclear. This study aims to clarify whether a preoperative lymphoscintigraphy is of additional benefit in a prospective randomized multicenter study design.

DETAILED DESCRIPTION:
Sentinel node biopsy is a well established tool for axillary staging in early breast cancer. So far the impact of a preoperative lymph node scintigraphy is unclear. Several studies indicate sentinel node biopsy to be a reliable method irrespective of prior lymph node scintigraphy, but data from prospective randomized trials are not available.

Although a preoperative lymph node scintigraphy is not explicitly demanded in current S3 guidelines in Germany its performance is a common practice.

If a preoperative lymphoscintigraphy could be safely omitted, possible benefits are a facilitation of the preoperative workflow as well as cost reduction for health care systems.

This study aims to clarify whether a preoperative lymphoscintigraphy is of additional benefit in a prospective randomized study design. In the two study arms sentinel node biopsy is performed either with or without knowledge of the preoperative lymphoscintigraphy findings. Primary end point is the average number of histologically detected sentinel lymph nodes per patient in both treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* invasive mamma carcinoma as verified by core cut biopsy
* extensive ductal carcinoma in situ as verified by core cut biopsy (at least 5 cm or at least 2,5 cm and G3 grading)
* clinical stage tumor T1-T3
* no signs of axillary lymph node metastasis on clinical examination including ultrasound examination
* no signs of distant metastatic disease
* male/ female patient in the age not less than 18 years
* Karnofsky performance status at least 70% or Eastern Cooperative Oncology Group (ECOG) score not higher than 1
* written patient informed consent

Exclusion Criteria:

* suspect axillary lymph nodes on clinical/ultrasound examination
* positive fine-needle biopsy of axillary lymph nodes
* sentinel lymph node biopsy to be performed after neoadjuvant chemotherapy
* recurrence of a mamma carcinoma
* prior extensive surgery of breast or axilla
* inflammatory or extramammary breast cancer
* pregnancy
* contraindication to the radionuclide
* inability to understand the studies purpose
* inability to receive surgery
* no written patient informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1198 (Actual)
Dates: Start 2014-05; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Average number of histologically detected sentinel lymph nodes per patient | Histological report expected within an average of 2 weeks after sentinel lymph node biopsy
  Number of resected sentinel lymph nodes is inversely correlated with false negative rate of sentinel lymph node biopsy. Average number of histologically detected sentinel lymph nodes per patient is assessed through pathologic report and serves as surrogate marker for false negative rate of sentinel node biopsy.

SECONDARY OUTCOMES:
Rate of patients with proven metastasis in sentinel lymph nodes | Histological report expected within an average of 2 weeks after sentinel lymph node biopsy
Rate of completion axillary dissection with proven metastasis in sentinel lymph nodes | histological report on subsequent completion axillary dissection within 6 months after initial sentinel lymph node biopsy
  A completion axillary dissection can be performed in case of proven metastasis in sentinel lymph nodes. A completion axillary dissection ca be performed either right away during sentinel lymph node biopsy or after completion of neoadjuvant chemotherapy. Hence assessment will be performed within 6 months after initial sentinel lymph node biopsy in order to include all patients planned for neoadjuvant chemotherapy.
Detection rates of sentinel nodes lymph nodes with preoperative lymphoscintigraphy vs. intraoperative gamma probe and histological detection rates of sentinel lymph nodes with vs. without preoperative access to lymphoscintigraphy | Histological report expected within an average of 2 weeks after sentinel lymph node biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Sherko Kümmel, MD, Principal Investigator — Kliniken Essen-Mitte; Thorsten Kühn, MD, Study Chair — Klinikum Esslingen; Johannes Holtschmidt, MD, Study Chair — Kliniken Essen-Mitte
Locations (23):
- Germany (22):
  - Kliniken Essen-Mitte, Essen, North Rhine-Westphalia
  - Brustzentrum im Klinikum Ansbach, Ansbach
  - Brustzentrum am Hochwaldkrankenhaus Bad Nauheim, Bad Nauheim
  - Kreisklinik Ebersberg, Brustzentrum, Ebersberg
  - Klinik für Frauenheilkunde & Geburtshilfe, Klinikum Esslingen, Esslingen am Neckar
  - Agaplesion Markus Krankenhaus Frankfurt, Brustzentrum, Frankfurt A. M.
  - Franziskus Hospital Harderberg, Brustzentrum Osnabrück, Georgsmarienhütte
  - Asklepios Harzkliniken Goslar, Brustzentrum, Goslar
  - Klinikum Gütersloh, Klinik für Frauenheilkunde und Geburtshilfe, Gütersloh
  - Sankt Elisabeth Krankenhaus Gütersloh, Frauenklinik, Gütersloh
  - Universitätsklinikum Hamburg Eppendorf, Hamburg
  - Kreiskrankenhaus Bergstrasse, Brustzentrum, Heppenheim an der Bergstrasse
  - Universitätsklinikum Schleswig-Holstein, Brustzentrum Kiel, Kiel
  - Universitätsfrauenklinik Magdeburg, Brustzentrum, Magdeburg
  - Evangelisches Krankenhaus Bethesda, Brustzentrum Niederrhein, Mönchengladbach
  - Universitätsfrauenklinik am Klinikum Südstadt Rostock, Rostock
  - DRK Krankenhaus Saarlouis, Brustzentrum, Saarlouis
  - Leopoldina Krankenhaus Schweinfurt, Brustzentrum, Schweinfurt
  - Klinikum St. Elisabeth Straubing, Brustzentrum, Straubing
  - Katharinen Hospital Unna, Brustzentrum, Unna
  - Kliniken Nordoberpfalz, Frauenklinik, Weiden
  - Marien-Hospital Wesel, Brustzentrum, Wesel
- Brustzentrum Bern, Engerriedspital/Lindenhofspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kuemmel S, Holtschmidt J, Gerber B, Von der Assen A, Heil J, Thill M, Krug D, Schem C, Denkert C, Lubitz J, Blohmer JU, Reinisch M, Hotzeldt M, Seither F, Nekljudova V, Schwidde I, Uhrhan K, Von Minckwitz G, Rezai M, Mulowski J, Loibl S, Kuehn T. Prospective, Multicenter, Randomized Phase III Trial Evaluating the Impact of Lymphoscintigraphy as Part of Sentinel Node Biopsy in Early Breast Cancer: SenSzi (GBG80) Trial. J Clin Oncol. 2019 Jun 10;37(17):1490-1498. doi: 10.1200/JCO.18.02092. Epub 2019 May 1. PMID 31042410
- [Result] Holtschmidt J, Kuemmel S, Krug D, Breit E, Kuehn T, Reinisch M. Reply to E. Hindie and A.K. Goel et al. J Clin Oncol. 2019 Oct 10;37(29):2705-2707. doi: 10.1200/JCO.19.01860. Epub 2019 Aug 29. No abstract available. PMID 31465263